CLINICAL TRIAL: NCT03138928
Title: XEN45 Gel Stent Implantation in Glaucoma Surgery
Brief Title: An Innovation in Glaucoma Surgery: XEN45 Gel Stent Implantation
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Sadık Altan Ozal, Ass. Proff, M.D., Trakya University
Other Study IDs: 14783785
Record Dates: First submitted 2017-04-25; First posted 2017-05-03 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Glaucoma Eye
Keywords: glaucoma; trabeculectomy; minimally invasive glaucoma surgery; XEN45 gel stent
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: XEN45 gel stent implantation in glaucoma surgery — The XEN gel stent (Allergan, Dublin, Ireland) is a recently developed, permanent, ab interno collagen implant that reduces IOP by draining aqueous fluid from the anterior chamber into the subconjunctival space

SUMMARY:
Purpose: To report the follow-up data for patients who had XEN45 gel stent implantation, a new method of minimally invasive glaucoma surgery (MIGS).

Material and Methods: Fifteen eyes of fifteen patients who had XEN45 gel stent implantation surgery were investigated in the study. All the patients were examined preoperatively and at the following postoperative time points: 1 day; 1 and 2 weeks; and 1, 2, 3, 6, and 12 months. Intraocular pressure (IOP) was measured by Goldmann applanation tonometry. Combined surgical procedures (XEN 45 + phacoemulsification + intraocular lens) were performed in the cases that had cataracts in addition to glaucoma.

DETAILED DESCRIPTION:
Introduction

Glaucoma is a group of eye diseases that results in damage to the optic nerve and permanent visual loss; more than 60 million people around the world are affected by glaucoma. Increased intraocular pressure (IOP) is the most important risk factor for the development of optic nerve damage and changes in the visual field. Therefore, the most effective treatment modality is the reduction of IOP, in order to prevent glaucoma progression and optic nerve atrophy. Trabeculectomy and episcleral aqueous drainage implants are currently the most widely used surgical methods for reducing IOP and treating glaucoma. Unfortunately, these procedures have potentially destructive intraoperative and postoperative complications, such as hypotony, choroidal effusion, blebitis, and endophthalmitis. Therefore, there is a trend of developing new surgical procedures to avoid the complications arising from conventional surgical procedures. These new surgical methods, called "minimally invasive glaucoma surgery" (MIGS), have some advantages over the conventional glaucoma surgical procedures, such as ab interno applicability, the elimination of external intervention requirements, and the ease of performance alongside cataract surgery. These advantages allow MIGS methods to be safer and less invasive than other surgical methods.

The XEN gel stent (Allergan, Dublin, Ireland) is a recently developed, permanent, ab interno collagen implant that reduces IOP by draining aqueous fluid from the anterior chamber into the subconjunctival space. The stent is a hydrophilic tube that is 6 mm long and composed of porcine gelatin crosslinked with glutaraldehyde. There are three sizes of this stent: 45 μm, 63 μm, and 140 μm, all with different inner diameters. The XEN45 gel stent is CE-marked in the European Union, and it is indicated for the treatment of refractory glaucoma that has proven resistant to previous surgical treatment and for patients with primary open angle glaucoma (POAG), pseudoexfoliative glaucoma, or pigmentary glaucoma that cannot be controlled with the maximum tolerated medical therapy. It is also licensed for use in Canada, Switzerland, and Turkey. The XEN45 gel stent was recently approved by the U.S. Food and Drug Administration (FDA). Because it is a new device, there are still unknown aspects of its efficacy and safety and of the proper surgical technique for its use. This study aimed to report the follow-up data after XEN45 gel stent implantation surgery in patients with different types of glaucoma.

Methods

This was a retrospective, consecutive case series study. Patients who had an XEN45 gel stent implantation surgery between January 2015 and March 2016 were enrolled in the study. Patients were included whose refractory glaucoma was resistant to previous surgical treatment. Patients were also included who had POAG, pseudoexfoliative glaucoma, or pigmentary glaucoma, with uncontrolled IOP and progressive visual field damage despite using the maximum tolerated dose of topical antiglaucomatous medications. Patients who had previous glaucoma surgery were included as well. The exclusion criteria included primary closed-angle glaucoma, a history of uveitis, and the presence of corneal disease. Patients who did not attend follow-up visits were also excluded. All patients were informed about the treatment and the potential complications. Informed patient consents were obtained preoperatively. The procedures of the study were approved by the institutional review board of the hospital and adhered to the tenets of the Declaration of Helsinki. The study protocol was approved by the local ethics committee (approval code: TUTF-BAEK 2016/213).

Before the XEN45 implantation, slit-lamp biomicroscopy and gonioscopic examination were performed. Intraocular pressure was measured by Goldmann applanation tonometry (AT 900, Haag Strait, Bern, Germany). A detailed fundus examination was done using a 78-dioptre non-contact lens after pupil dilatation by 1% tropicamide gutt.

All of the surgical procedures were performed under sterile conditions by the same surgeon (OK). Irrigation of the eyelashes, eyelids, and periorbicular tissues was performed with antiseptic 10% povidone iodine. While using an eye speculum, 5% povidone iodine was flushed onto the conjunctiva and fornix for two minutes; conjunctival irrigation was then completed with saline. The surgery was performed under peribulbar anaesthesia with 5 mL prilocaine and 5 mL bupivacaine. After peribulbar anaesthesia, the superonasal quadrant of the conjunctiva was marked by blue surgical dye 3 mm posterior to the limbus. Clear corneal incisions (main and side-port) were created in the inferotemporal and superotemporal quadrants; a highly cohesive viscoelastic was used to stabilise the anterior chamber during surgery. A 27-gauge pre-loaded injector was placed into the eye through the main clear corneal incision at the inferotemporal quadrant. The needle was directed toward the superonasal quadrant (Figure 3). One hand was used to manipulate the injector, and the other hand was used to fix and rotate the eye. The needle was pushed into the sclera and carried forward into the subconjunctival space. The surgery was performed under gonioscopic control. A 6-mm-long implant was created to be positioned 2 mm into the subconjunctival space, 3 mm into the sclera, and 1 mm into the anterior chamber. Therefore, visualization of the tip of the needle exiting from the sclera indicated that an optimal 3-mm intrascleral tunnel had been formed. The XEN45 implant was deployed by rotating a dial on the inserter. Once bleb formation was seen, the needle was withdrawn. The viscoelastic material was aspirated, and then 0.1 ml of 1% cefuroxime was injected into the anterior chamber. Finally, the clear corneal incisions were hydrated with a balanced salt solution. Mitomycin C was not injected into the conjunctiva at any stage of the surgery. Topical steroid and antibiotic treatments were applied after the surgery. A topical steroid (prednisolone acetate 1%) was applied six or more times daily to control postoperative intraocular inflammation. The topical steroid treatment was stopped after the first month postoperative. Ocular massage for one minute four times daily was recommended during the postoperative period. Needling was not performed at any of the postoperative visits. Topical antiglaucomatous medications were added as needed according to the postoperative IOP levels. Follow-up visits were planned for 1 day, 1 and 2 weeks, and 1, 2, 3, 6, and 12 months.

Combined surgery (XEN45 + phacoemulsification + intraocular lens) was performed in the cases that had cataracts in addition to glaucoma. In combined surgery, the XEN45 implantation was performed after the phacoemulsification. After the intraocular lens implantation in the capsular sac, the anterior chamber was filled with a highly cohesive viscoelastic material. Then, the same procedures as were described previously were carried out.

All the data were compiled into a computer file for statistical analysis, and Statistical Package for Social Sciences for Windows 17.0 was used to perform the Wilcoxon signed ranks test. A p value less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Primary open-angle glaucoma, pseudoexfoliative glaucoma, or pigmentary glaucoma, with uncontrolled IOP and progressive visual field damage despite using the maximum tolerated dose of topical antiglaucomatous medications. Patients who had previous glaucoma surgery were included as well.

Exclusion Criteria:

* The exclusion criteria included primary closed-angle glaucoma, a history of uveitis, and the presence of corneal disease. Patients who did not attend follow-up visits were also excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifteen patients who had an XEN45 gel stent implantation surgery between January 2015 and March 2016 were enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | Postoperative 12 months
  Mean intraocular pressure values

SECONDARY OUTCOMES:
Antiglaucomatous medications | Postoperative 12 months
  Mean number of antiglaucomatous medications
Incidence of complications | Postoperative 12 months
  Complications due to surgery

IPD SHARING:
Plan to Share IPD: Yes
This clinical trial is under review for publishing. If it is accepted for publishing,our results will be shared.

REFERENCES:
- [Background] Sheybani A, Lenzhofer M, Hohensinn M, Reitsamer H, Ahmed II. Phacoemulsification combined with a new ab interno gel stent to treat open-angle glaucoma: Pilot study. J Cataract Refract Surg. 2015 Sep;41(9):1905-9. doi: 10.1016/j.jcrs.2015.01.019. Epub 2015 Oct 23. PMID 26482822
- [Result] Tham YC, Li X, Wong TY, Quigley HA, Aung T, Cheng CY. Global prevalence of glaucoma and projections of glaucoma burden through 2040: a systematic review and meta-analysis. Ophthalmology. 2014 Nov;121(11):2081-90. doi: 10.1016/j.ophtha.2014.05.013. Epub 2014 Jun 26. PMID 24974815
- [Result] Heijl A, Leske MC, Bengtsson B, Hyman L, Bengtsson B, Hussein M; Early Manifest Glaucoma Trial Group. Reduction of intraocular pressure and glaucoma progression: results from the Early Manifest Glaucoma Trial. Arch Ophthalmol. 2002 Oct;120(10):1268-79. doi: 10.1001/archopht.120.10.1268. PMID 12365904
- [Result] Nouri-Mahdavi K, Brigatti L, Weitzman M, Caprioli J. Outcomes of trabeculectomy for primary open-angle glaucoma. Ophthalmology. 1995 Dec;102(12):1760-9. doi: 10.1016/s0161-6420(95)30796-8. PMID 9098275
- [Result] Landers J, Martin K, Sarkies N, Bourne R, Watson P. A twenty-year follow-up study of trabeculectomy: risk factors and outcomes. Ophthalmology. 2012 Apr;119(4):694-702. doi: 10.1016/j.ophtha.2011.09.043. Epub 2011 Dec 23. PMID 22196977
- [Result] Minckler D, Mosaed S, Dustin L, Ms BF; Trabectome Study Group. Trabectome (trabeculectomy-internal approach): additional experience and extended follow-up. Trans Am Ophthalmol Soc. 2008;106:149-59; discussion 159-60. PMID 19277230
- [Result] Ting JL, Damji KF, Stiles MC; Trabectome Study Group. Ab interno trabeculectomy: outcomes in exfoliation versus primary open-angle glaucoma. J Cataract Refract Surg. 2012 Feb;38(2):315-23. doi: 10.1016/j.jcrs.2011.08.043. PMID 22322166
- [Result] Bussel II, Kaplowitz K, Schuman JS, Loewen NA; Trabectome Study Group. Outcomes of ab interno trabeculectomy with the trabectome by degree of angle opening. Br J Ophthalmol. 2015 Jul;99(7):914-9. doi: 10.1136/bjophthalmol-2014-305577. Epub 2014 Oct 21. PMID 25336577
- [Result] Lewis RA. Ab interno approach to the subconjunctival space using a collagen glaucoma stent. J Cataract Refract Surg. 2014 Aug;40(8):1301-6. doi: 10.1016/j.jcrs.2014.01.032. Epub 2014 Jun 15. PMID 24943904
- [Result] Vera V, Horvath C. Xen Gel Stent: The solution designed by AqueSys. In: Samples, JR, Ahmed, IIK, editors. Surgical innovations in glaucoma. New York: Springer Science+Business Media; 2014, p. 189-198.
- [Result] Richter GM, Coleman AL. Minimally invasive glaucoma surgery: current status and future prospects. Clin Ophthalmol. 2016 Jan 28;10:189-206. doi: 10.2147/OPTH.S80490. eCollection 2016. PMID 26869753
- [Result] Kerr NM, Wang J, Barton K. Minimally invasive glaucoma surgery as primary stand-alone surgery for glaucoma. Clin Exp Ophthalmol. 2017 May;45(4):393-400. doi: 10.1111/ceo.12888. Epub 2017 Jan 29. PMID 27928879
- [Result] Garcia-Feijoo J, Sampaolesi JR. A multicenter evaluation of ocular surface disease prevalence in patients with glaucoma. Clin Ophthalmol. 2012;6:441-6. doi: 10.2147/OPTH.S29158. Epub 2012 Mar 22. PMID 22536034
- [Result] Valente C, Iester M, Corsi E, Rolando M. Symptoms and signs of tear film dysfunction in glaucomatous patients. J Ocul Pharmacol Ther. 2011 Jun;27(3):281-5. doi: 10.1089/jop.2010.0133. Epub 2011 May 10. PMID 21557633
- [Result] Dupont G, Collignon N. [NEW SURGICAL APPROACH IN PRIMARY OPEN-ANGLE GLAUCOMA: XEN GEL STENT A MINIMALLY INVASIVE TECHNIQUE]. Rev Med Liege. 2016 Feb;71(2):90-3. French. PMID 27141652
- [Result] Perez-Torregrosa VT, Olate-Perez A, Cerda-Ibanez M, Gargallo-Benedicto A, Osorio-Alayo V, Barreiro-Rego A, Duch-Samper A. Combined phacoemulsification and XEN45 surgery from a temporal approach and 2 incisions. Arch Soc Esp Oftalmol. 2016 Sep;91(9):415-21. doi: 10.1016/j.oftal.2016.02.006. Epub 2016 Mar 16. English, Spanish. PMID 26995503
- [Result] Pinto Ferreira N, Abegao Pinto L, Marques-Neves C. XEN Gel Stent Internal Ostium Occlusion: Ab-Interno Revision. J Glaucoma. 2017 Apr;26(4):e150-e152. doi: 10.1097/IJG.0000000000000625. PMID 28098579